CLINICAL TRIAL: NCT00639717
Title: Addition of Etanercept and Extracorporeal Photopheresis to Standard GVHD Prophylaxis in Patients Undergoing Reduced Intensity Unrelated Donor Hematopoietic Stem Cell Transplant
Brief Title: Addition of Etanercept and Extracorporeal Photopheresis (ECP) to Standard Graft-Versus-Host Disease (GVHD) Prophylaxis in Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Mallinckrodt (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: umcc 2008.003
Record Dates: First submitted 2008-03-11; First posted 2008-03-20 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Graft Versus Host Disease
Keywords: GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid; Etanercept; Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept and ECP (Experimental): Etanercept and ECP (Extracorporeal Photopheresis) in addition to standard GVHD prevention:
  Etanercept will be given twice weekly by subcutaneous injection starting on the day of HSCT (Hematopoietic stem cell transplantation) conditioning until 8 weeks post transplant. ECP treatments will begin at once weekly starting at 4 weeks post transplant and continue at less frequent intervals until 6 months post transplant.
  GVHD prophylaxis will consist of a standard two drug regimen: mycophenolate for 4 weeks and tacrolimus (titrated to a therapeutic level) for 8 weeks, then weaned over 4 months with discontinuation by 6 months post-transplant.
  Interventions: Procedure: stem cell transplant; Drug: tacrolimus (standard GVHD prophylaxis); Drug: mycophenolate (standard GVHD prophylaxis); Drug: etanercept; Drug: methoxsalen

INTERVENTIONS:
Procedure: stem cell transplant — reduced intensity, matched unrelated donor stem cell transplant
Drug: tacrolimus (standard GVHD prophylaxis) — Tacrolimus(or cyclosporine when necessary)
  Tacrolimus will begin on day -3, IV or oral.
  Target trough level for tacrolimus is 8-12 ng/ml.
  In the absence of GVHD, tacrolimus tapering will begin on day +56 post transplant
Drug: mycophenolate (standard GVHD prophylaxis) — Mycophenolate will begin on day 0 at 10 mg/kg/dose (up to 1 gram per dose) every 8 hours orally or intravenously and will continue until day 28.
Drug: etanercept — Etanercept will be given at a dose 0.4 mg/kg (actual weight) up to a maximum dose of 25 mg, subcutaneously, twice weekly from day 0 to day 56 (16 doses)
  Other Names: Enbrel
Drug: methoxsalen — Methoxsalen (UVADEX) treatments by Extracorporeal photopheresis (ECP) will be started day +28 post transplant and given weekly.
  On day +70 post transplant ECP frequency will be given every other week.
  On day +100 post transplant ECP will be given monthly until day +180 and stopped.
  Other Names: UVADEX

SUMMARY:
This research study investigates the benefits and possible risks of adding both etanercept (Enbrel) and ECP (extracorporeal photopheresis) to the conventional preventative (or prophylactic) treatments for graft-versus-host disease (GVHD). GVHD is a common, serious, and too often fatal, complication after matched unrelated donor stem cell transplantation, regardless of the pre-transplant conditioning regimen used (full or reduced intensity).

Reduced intensity transplants which employ lower doses of chemotherapy during the conditioning phase of the transplant, are less toxic than full intensity transplants. Reduced intensity transplants may extend the unrelated donor transplant option to older patients or to patients with existing medical conditions or illness, where a full intensity transplant is not possible. To be successful, reduced intensity transplants need to offset any lower effectiveness in killing cancer cells during the conditioning phase, with the establishment of a donor cell, graft-versus-leukemia effect (GVL). The GVL effect and GVHD are associated with each other and therefore, the goal of GVHD prophylaxis for this study is not so much to prevent all GVHD, but rather to prevent serious and fatal acute GVHD.

Most GVHD-related deaths are either the direct consequence of severe GVHD or from infections associated with intense immunosuppression, a consequence of the standard treatments for acute GVHD, which almost always include high-dose steroids. A more effective prophylaxis therapy that allows for the GVL effect to develop, while limiting the exposure to high-dose steroids may reduce transplant mortality and morbidity. We also will study how key chemical and cellular factors relate to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for unrelated donor (allogeneic) HSCT for hematologic conditions, either malignant or non-malignant.
* Donor can be unrelated marrow, blood or cord blood.
* Any disease for which unrelated donor transplant is appropriate is eligible except:

  * Progressive or poorly controlled malignancies for which the likelihood of durable disease control [i.e., patients expected to have at least 6 months PFS from date of transplant] is <25%.
  * This determination of likelihood of durable disease control must take into account the patient's disease status and consideration of the agents and doses used in the reduced intensity conditioning regimen.
  * The determination of adequate disease control will be certified by the PI or designee on the eligibility checklist.
  * Patients may be consented to this trial based on disease control at the time of consent, but later removed from the trial prior to initiation of transplant conditioning regimen if disease status confirmation between consenting and transplant changes. In the event this occurs these patients will be replaced.
* Must be receiving a recognized reduced intensity transplant as determined by the University of Michigan Blood and Marrow Transplantation Program.
* Patients age 50 or older are eligible based on age.
* Patients may be <50 years old if they are eligible for a reduced intensity conditioning regimen based on disease type (eg, indolent lymphoma) or if comorbidities preclude a full-intensity transplant.
* Patients must have adequate venous access by either peripheral vein or central line so that ECP can be performed.
* Patients must be expected to tolerate the fluid shifts associated with ECP. The primary reason for expected intolerance of ECP is small size (ie, <30kg weight), but other factors may also be considered in this determination.

Exclusion Criteria:

* Not a candidate for a reduced intensity transplant conditioning regimen (based on the current U-M BMT program clinical guidelines).
* Patient has a suitable related donor available for transplant.
* Karnofsky or Lansky performance status of < 50% at the time of admission for HSCT
* Patients with evidence of HIV infection or other opportunistic infection including but not limited to Tuberculosis and Histoplasmosis.
* Patients with active bacterial, fungal or viral infection not responding to treatment.
* Any medical or psychological conditions that would keep the patient from complying with the protocol and/or would markedly increase the morbidity and mortality from the procedure.
* Pregnancy.
* T-cell depleted allograft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Yanik, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept and ECP: Etanercept and ECP (Extracorporeal Photopheresis) in addition to standard GVHD prevention:
  Etanercept will be given twice weekly by subcutaneous injection starting on the day of HSCT conditioning until 8 weeks post transplant. ECP treatments will begin at once weekly starting at 4 weeks post transplant and continue at less frequent intervals until 6 months post transplant.
  GVHD prophylaxis will consist of a standard two drug regimen: mycophenolate for 4 weeks and tacrolimus (titrated to a therapeutic level) for 8 weeks, then weaned over 4 months with discontinuation by 6 months post-transplant.
Period: Overall Study
Arm/Group | Etanercept and ECP
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 60 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive at 6 Months
Description: Overall survival at 6 months
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 48
percentage of patients | 83 [73 to 95]

2. Primary Outcome: Percentage of Patients Who Experienced Relapse by 6 Months
Description: Relapse rate at 6 months. Relapse is defined as recurrence of disease.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 48
Percentage of patients | 8 [0 to 16]

3. Secondary Outcome: The Percentage of Patients That Experienced Graft Versus Host Disease
Description: Incidence of acute GVHD grades 2-4 and chronic GVHD in this study population
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 48
percentage of patients | 46 [32 to 60]

4. Secondary Outcome: Measured Level of Circulating Plasma Markers After Transplant
Time Frame: 100 days
Population: Plasma markers were not analyzed.
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 0

5. Secondary Outcome: Regulatory T Cell Numbers Post-transplant
Time Frame: 180 days
Population: T cell numbers were not analyzed
Arm/Group | Etanercept and ECP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Etanercept and ECP
Serious Adverse Events (participants affected / at risk) | 19/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept and ECP (N=48)
Blood Bone Marrow - Other (Blood and lymphatic system disorders) | 3 (3)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1)
Ileus, GI Obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Vascular disorders) | 1 (1)
Hemorrhage, GI (Vascular disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Stomach Infection (Infections and infestations) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Pain - Cardiac (Cardiac disorders) | 1 (1)
Pain - Head (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept and ECP (N=48)
Blood Bone Marrow - Other (Blood and lymphatic system disorders) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Cardiac ischemia/infarction (Cardiac disorders) | 4 (4)
Hypertension (Cardiac disorders) | 4 (5)
PTT (Partial Thromboplastin Time) (Vascular disorders) | 4 (6)
Ascites (non-malignant) (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 12 (13)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 4 (6)
Febrile neutropenia (Infections and infestations) | 13 (13)
Blood Infection with Grade 3/4 ANC (Infections and infestations) | 9 (10)
Lung Infection (Infections and infestations) | 5 (6)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Blood Infection with Normal ANC (Infections and infestations) | 8 (8)
Catheter-related Infection (Infections and infestations) | 4 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 (5)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (4)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 (6)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (6)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 17 (35)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 11 (18)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 9 (11)
Muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 3 (3)
Ataxia (incoordination) (Nervous system disorders) | 6 (11)
Confusion (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 3 (3)
Anxiety (Nervous system disorders) | 3 (3)
Somnolence/depressed level of consciousness (Nervous system disorders) | 5 (6)
Pain-Abdomen (Gastrointestinal disorders) | 4 (5)
Pain-Back (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain-Head (Nervous system disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes